CLINICAL TRIAL: NCT05933824
Title: A Randomized, Placebo-controlled, Single-administration, Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of LP-98 Injection in Healthy Subjects in a First-in-human Clinical Study
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of LP-98 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanxi Kangbao Biological Product Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KB_LP-98_101
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2023-12

CONDITIONS: Hiv
Keywords: Healthy Subjects; safety and tolerability; pharmacokinetic (PK); immunogenicity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- PartA:Dose level(5mg) (Experimental): Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
  Interventions: Drug: LP-98 injection
- PartA:Dose level(10mg) (Experimental): Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
  Interventions: Drug: LP-98 injection
- PartA:Dose level(20mg) (Experimental): Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
  Interventions: Drug: LP-98 injection
- PartA:Dose level(40mg) (Experimental): Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
  Interventions: Drug: LP-98 injection
- PartA:Dose level(80mg) (Experimental): Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(5mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(10mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(20mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(40mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(80mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection
- PartB:Dose level(160mg) (Experimental): Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.
  Interventions: Drug: LP-98 injection

INTERVENTIONS:
Drug: LP-98 injection — Part A is administration is by subcutaneous LP98/placebo,Part B is administration is by intravenous drip LP98/placebo
  Other Names: placebo-controlled

SUMMARY:
A randomized, placebo-controlled, single-administration, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of LP-98 injection in healthy subjects in a first-in-human clinical study

DETAILED DESCRIPTION:
The study was divided into two parts, Part A and Part B. The Part A and Part B studies were carried out separately according to the protocol flow, with the Part A study carried out first.

1. Part A is set up with 5 cohorts(5mg, 10mg, 20mg, 40mg, 80mg), administration is by subcutaneous, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 5, to observe the safety, tolerability, PK and ADA of LP-98 injection by subcutaneous.
2. Part B is set up with 6 cohorts (5mg,10mg,20mg,40mg,80mg, 160mg), administration is by intravenous drip, each subject entered only one cohort to receive the drug. 4 subjects were included in cohort 1, and 8 subjects were planned to be included in each cohort 2 to 6, to observe the safety, tolerability, PK and ADA of LP-98 injection by intravenous drip.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria for study entry:

1. Willing to participate in the study and sign ICF with clear date;
2. Aged 18 to 55 years at the screening visit, male or female;
3. Body weight ≥ 50 kg for males or body weight ≥ 45 kg for females, and body mass index (BMI) within the range of 19 to 28 kg/m2 (inclusive);
4. Be in good health in the PI's judgment, with no clinical significance in previous medical history, laboratory tests, physical examinations, vital signs, and ECG findings;
5. All subjects and his/her partners must agree to use effective non-drug contraception (except for subjects had permanent contraception, i.e., bilateral tubal ligation or vasectomy, etc.) from 2 weeks prior to screening to 3 months after finishing the study. Females must have a negative serum human chorionic gonadotropin (hCG) test for pregnancy confirmation at screening;
6. Willing to comply with the visits, treatments, laboratory tests and other study process required by the protocol.

Exclusion Criteria:

1. Allergic to the IP or its excipients, or medicine of the same class , or having a history of severe allergies (including any food allergy or drug allergy);
2. With history or family history of psychiatric, or history of chronic or serious disorders of the central nervous system, cardiovascular, hepatic, nephrological, pulmanory, digestive, metabolic, hematological or skeletal system etc., or definitive history of myelosuppression, orany other significant history of disease that may affect the safety or PK parameters in the PI's judgment;
3. Having positive result for human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or Treponema pallidum antibody;
4. Having clinically significant abnormal results of vital signs or laboratory tests required by the protocol;
5. Having clinically significant abnormality of 12-lead ECG, or having a QTcF interval (using Fridericia's correction) > 450 ms for males or > 470 ms for females;
6. With serum creatine clearance rate (Ccr) < 80 ml/min/1.73 m2 (based on Cockcroft-Gault formula);
7. Known or suspected history of drug abuse (i.e., morphine, methamphetamine, ketamine, dimethylenedioxymethamphetamine, tetrahydrocannabinol acid, cocaine etc.), or having positive result for drug abuse;
8. With history of heavy alcohol consumption within 1 year prior to screening (more than 21 units of alcohol per week, i.e., 360 ml of 5% beer, 45 ml of 40% hard liquor, 120 ml of 12% wine, or positive alcohol test;
9. Smoking more than 5 cigarettes per day within 3 months prior to screening, or inability to comply with the prohibition of smoking during the study;
10. Consuming amount > 6 servings of coffee, tea, cola, energy-drink, or other caffeine-containing product per day. One serving ≈ 120 mg of caffeine. Or consumed any caffeine-containing product within 24 hours prior to the dosing of the IP;
11. Had received vaccination within 30 days prior to screening, or planning to receive vaccination during the study;
12. Had received any prescription and non-prescription drugs, herbal remedies, or dietary supplements within 14 days prior to the dosing of the IP;
13. Participated in any other clinical trial within 3 months prior to screening;
14. Had received surgical operation within 3 months prior to screening, or planning to receive surgical operation during the study;
15. Currently pregnant or lactating women；
16. Had blood donation or blood loss over 200 mL within 3 months prior to screening, or planning to donate blood during the study；
17. Cannot tolerate venipuncture blood collection and/or have a history of blood or needle sickness
18. Other conditions considered to be ineligible for study entry in the PI's judgment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in respiration rate of Vital Signs | Within 36 days after the first administration.
  Respiration rate in times / minute
Changes from baseline in blood pressure of Vital Signs. | Within 36 days after the first administration.
  Blood pressure in mmHg
Changes from baseline in body temperature of Vital Signs. | Within 36 days after the first administration.
  Body temperature in Celsius degree
Changes from baseline in ECG PR intervalThe cardiac rhythm is showed in 12 Leads | within 36 days after administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG QRS intervalThe cardiac rhythm is showed in 12 Leads | within 36 days after administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG QT intervalThe cardiac rhythm is showed in 12 Leads | within 36 days after administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in Blood lactate of Laboratory Examination. | within 36 days after administration
  Changes of blood lactate will be recorded.
Changes from baseline in Pregnancy test of Laboratory Examination. | within 36 days after administration
  Pregnancy test will be tested in female subjects.
Changes from baseline in red blood cell count of Laboratory Examination. | within 36 days after administration
  Red blood cell count in whole blood is reported in the form of number.
Changes from baseline in white blood cell count of Laboratory Examination. | within 36 days after administration
  White blood cell count in whole blood is reported in the form of number.
Changes from baseline in neutrophil count of Laboratory Examination. | within 36 days after administration
  Neutrophil count in whole blood is reported in the form of number.
Changes from baseline in lymphocyte count of Laboratory Examination. | within 36 days after administration
  Lymphocyte count in whole blood is reported in the form of number.
Changes from baseline in platelet count of Laboratory Examination. | within 36 days after administration
  Platelet count in whole blood is reported in the form of number.
Changes from baseline in hemoglobin of Laboratory Examination. | within 36 days after administration
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination. | within 36 days after administration
  Prothrombin time (PT) is a screening test for exogenous coagulation factors.
Changes from baseline in INR of Laboratory Examination. | within 36 days after administration
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent.
Changes from baseline in APTT of Laboratory Examination. | within 36 days after administration
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in direct bilirubin of Laboratory Examination. | within 36 days after administration
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in ALT of Laboratory Examination. | within 36 days after administration
  Changes of ALT concentration (U/L) in serum will be recorded.
Changes from baseline in AST of Laboratory Examination. | within 36 days after administration
  Changes of AST concentration (U/L) in serum will be recorded.
Changes from baseline in total protein of Laboratory Examination. | within 36 days after administration
  Changes of total protein concentration (g/L) in serum will be recorded.
Changes from baseline in albumin of Laboratory Examination. | within 36 days after administration
  Changes of albumin concentration (g/L) in serum will be recorded.
Changes from baseline in creatinine of Laboratory Examination. | within 36 days after administration
  Changes of creatinine concentration (μmol/L) in serum will be recorded.
Changes from baseline in glucose of Laboratory Examination | within 36 days after administration
  Changes of glucose concentration (mmol/L) in serum will be recorded.
Changes from baseline in potassium of Laboratory Examination. | within 36 days after administration
  Changes of potassium concentration (mmol/L) in serum will be recorded.
Changes from baseline in sodium of Laboratory Examination. | within 36 days after administration
  Changes of sodium concentration (mmol/L) in serum will be recorded.
Changes from baseline in chlorine of Laboratory Examination. | within 36 days after administration
  Changes of chlorine concentration (mmol/L) in serum will be recorded.
Changes from baseline in urine specific gravity of Laboratory Examination. | within 36 days after administration
  Changes of urine specific gravity will be recorded.
Changes from baseline in urine pH of Laboratory Examination. | within 36 days after administration
  Changes of urine pH value will be recorded.
Changes from baseline in urine glucose of Laboratory Examination. | within 36 days after administration
  Changes of urine glucose will be examined by qualitative test (positive or negative).
Changes from baseline in urine protein of Laboratory Examination. | within 36 days after administration
  Changes of urine protein will be examined by qualitative test (positive or negative).
Changes from baseline in urine ketone body of Laboratory Examination. | within 36 days after administration
  Changes of urine ketone body will be examined by qualitative test (positive or negative).
Changes from baseline in urine white blood cell of Laboratory Examination. | within 36 days after administration
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative).
Changes from baseline in urine occult blood of Laboratory Examination. | within 36 days after administration
  Changes of urine occult blood will be examined by qualitative test (positive or negative).
Changes from baseline in CK of Laboratory Examination | within 36 days after administration
  Changes of CK concentration (U/L) in serum will be recorded.
Changes from baseline in CK-MB of Laboratory Examination | within 36 days after administration
  Changes of CK-MB concentration (ng/mL) in serum will be recorded.
Changes from baseline in LDH of Laboratory Examination | within 36 days after administration
  Changes of LDH concentration (U/L) in serum will be recorded.
Changes from baseline in ALP of Laboratory Examination | within 36 days after administration
  Changes of ALP concentration (U/L) in serum will be recorded.
Changes from baseline in Triglyceride of Laboratory Examination | within 36 days after administration
  Changes of Triglyceride concentration (mmol/L) in serum will be recorded.
Changes from baseline in CHOL of Laboratory Examination | within 36 days after administration
  Changes of CHOL concentration (mmol/L) in serum will be recorded.

SECONDARY OUTCOMES:
Changes from baseline in Immunogenic blood collection of Laboratory Examination. | within 36 days after administration
  Changes of immunogenic blood collection will be recorded.The historical changes of test results (including positive rate and titer) of various indicators were counted.
Pharmacokinetics：Cmax | within 36 days after administration
  pharmacokinetic characteristics of Lipovirtide in infected patients：Cmax
Pharmacokinetics：AUC0-t | within 36 days after administration
  pharmacokinetic characteristics of Lipovirtide in infected patients：AUC0-t
Pharmacokinetics：AUC0-∞ | within 36 days after administration
  pharmacokinetic characteristics of Lipovirtide in infected patients：AUC0-∞

OTHER OUTCOMES:
Explore changes in biomarkers (CD4+, CD8+T cell counts) from baseline after administration | within 36 days after administration
  Changes of CD4+T cell counts will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, Master, Principal Investigator — Henan Provincial Hospital for Infectious Diseases (Zhengzhou Sixth People's Hospital)
Locations (1):
- Henan Provincial Hospital for Infectious Diseases (Zhengzhou Sixth People's Hospital), Zhengzhou, Henan, China